CLINICAL TRIAL: NCT07066332
Title: The Use of Cornell Note Taking as a Teaching Technique in Nursing Education: A Randomised Controlled Study
Brief Title: Effect of Cornell Note Taking as a Teaching Techinique in Nursing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Nadiye BARIŞ EREN, Asst. Prof., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TarsusU-NBARISEREN-004
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Education Nursing
Keywords: motivation; listening skills; Note taking; education; nursing students

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cornell Note Taking education group (Experimental): In the first stage, students will be informed about the research and their consent will be obtained. The 'Personal Information Form' will be filled in under observation in the classroom environment by the students whose informed consent is obtained and who agree to participate in the research. Then, 'Achievement Test 1' and 'Motivation Scale for Instructional Material' and 'Listening Skill Scale' will be applied to all students as pre-test. In the second stage, Cornell note-taking technique training will be given. In the third stage, Cornell note-taking technique templates will be distributed and they will be asked to fill them in the scope of the subject of Excretory activities in line with the training they have received. In the fourth stage, the subject of Excretory activities will be explained to the intervention and control groups separately. In the fifth stage, one week after the training, 'Achievement Test 2' and 'Motivation Scale for Teaching Material' and 'Listening Skill Sca
  Interventions: Behavioral: Cornell Note Taking education group
- Control Group (No Intervention): In the first stage, students will be informed about the research and their consent will be obtained. The 'Personal Information Form' will be filled in under observation in the classroom environment by the students whose informed consent is obtained and who agree to participate in the research. Then, 'Achievement Test 1' and 'Motivation Scale for Instructional Material' and 'Listening Skill Scale' will be applied to all students as pre-test. In the second stage, no intervention will be made to the control group. In the third stage, routine lecturing will be continued without any intervention to the control group. In the fourth stage, the subject of Excretory activities will be explained to the intervention and control groups separately. In the fifth stage, one week after the training, 'Achievement Test 2' and 'Motivation Scale for Teaching Material' and 'Listening Skill Scale' will be applied to the students as a post-test.

INTERVENTIONS:
Behavioral: Cornell Note Taking education group — Students will be trained in the Cornell note-taking technique.
  Arms: Cornell Note Taking education group

SUMMARY:
This study was conducted to evaluate the effect of Cornell note-taking technique on knowledge level, learning motivation and listening skills in nursing students.

Research hypotheses:

H1. Using the Cornell note-taking technique increases the academic success of nursing students.

H2. Using the Cornell note-taking technique increases the motivation of nursing students.

H3. Using the Cornell note-taking technique increases the listening skills of nursing students.

DETAILED DESCRIPTION:
Note-taking is part of the learning process. Students take short notes in a way that they will remember later in the lesson. It was observed that students who took short reminder notes achieved more successful results than students who took detailed notes. In the same way, the rate of remembering the subject matter of the students who took notes was approximately 2 times higher than those who did not take notes. In another study, note-taking skills ranked second among the skills that students need to improve. There are studies showing that note-taking improves academic performance. For this, it is also necessary for students to improve their listening skills. Although studies have revealed that Cornell note-taking technique has positive effects, there are very limited studies in the literature on the use of Cornell note-taking technique in nursing students. This study was planned to evaluate the effect of Cornell note-taking technique on knowledge level, learning motivation and listening skills in nursing students. It is thought that Cornell note-taking technique can be used for all nursing students and can make the learning process more enjoyable, increase participation in lessons, increase motivation, and positively affect the level of listening and success.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being 18 years of age or older
* Being a first year student
* Taking the Fundamentals of Nursing course for the first time
* Not being a student who came via horizontal or vertical transfer
* Not having received training on 'Excretory Activities'
* Not having been absent on the dates when the research data will be collected

Exclusion Criteria:

* Not volunteering to participate in the research
* Being under 18 years old
* Not being a first year student
* Being a student who came via horizontal or vertical transfer
* Being a health vocational high school graduate
* Being a student in the intervention group who did not attend the Cornell note-taking technique training
* Being a student in the control group who found to have reached the Cornell note-taking technique template

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | 10 minutes
  This form was prepared by the researchers in line with the literature and includes questions questioning the demographic characteristics of the students such as age, gender, socioeconomic level, etc. This form will be used before the training.
Achievement Test 1 | 20 minutes
  It consists of 25 multiple choice questions on the topic of "Excretory activities". This form will be used before the training.
Motivation Scale for Instructional Material | 10 minutes
  It will be used to measure motivations regarding instructional material. The scale is a 33-item, 5-point Likert type. The highest score that can be obtained from the entire scale is 165, and the lowest score is 33. This form will be used before and after the training.
Listening Skill Scale | 10 minutes
  It will be used to measure students' listening skills. The scale is a 15-item 5-point Likert type. The highest score that can be obtained from the entire scale is 75, the lowest score is 15. This form will be used before and after the training.
Achievement Test 2 | 20 minutes
  It consists of 25 multiple choice questions on the topic of "Excretory activities". This form will be used after the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No